CLINICAL TRIAL: NCT05046431
Title: A Multicenter, Double-blind, Randomized, Parallel-group Study to Compare the Efficacy and Safety of BAT2506 Versus Simponi® in Participants With Active Psoriatic Arthritis
Brief Title: Comparative Study of BAT2506 With Simponi® in Participants With Active Psoriatic Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAT-2506-002-CR
Record Dates: First submitted 2021-09-13; First posted 2021-09-16 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EU Simponi (Active Comparator)
  Interventions: Drug: EU Simponi
- BAT2506 (Experimental)
  Interventions: Drug: BAT2506

INTERVENTIONS:
Drug: BAT2506 — 50mg/0.5mL
  Arms: BAT2506
Drug: EU Simponi — 50mg/0.5mL
  Arms: EU Simponi

SUMMARY:
This is a multicenter, double-blind, randomized, parallel-group study to compare the efficacy,pharmacodynamics (PD), pharmacokinetics (PK), safety, and immunogenicity of BAT2506 versus Simponi® in participants with active PsA.

The study will consist of up to 4-week Screening Period, a 52-week Treatment Period, and a 8-week Safety Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

* Participant has PsA for at least 6 months prior to the first administration of the study drug and meets classification criteria for PsA (CASPAR) at Screening.
* Participant has active PsA defined by the presence of ≥3 of 68 tender joint counts and ≥3 of 66 swollen joint counts at Screening and Randomization.
* Participant has active PsA at Screening despite previous DMARD or NSAID therapy. DMARD therapy is defined as taking DMARD for at least 3 months, or evidence of DMARD intolerance. NSAID therapy is defined as taking an NSAID for at least 4 weeks (or have intolerance to or contraindication to NSAID therapy).
* Participant has at least 1 active psoriatic lesion with a qualifying lesion of at least 2 cm in diameter at Screening and Randomization.
* Participant is negative for rheumatoid factor and anti-cyclic citrullinated peptide (ACCP) antibodies at Screening.

Exclusion Criteria:

* Participant is currently receiving or has previously received any biological agent or targeted disease modifying anti-rheumatic drugs (DMARDs) for the treatment of PsA or psoriasis.
* Participant has previously received any other nonbiological DMARDs (apart from MTX), including sulfasalazine, hydroxychloroquine or apremilast within 8 weeks prior to the first administration of the study drug; or has previously received leflunomide within 12 weeks (except at least 4 weeks prior to the first administration of the study drug, the subject has documented completion of standard cholestyramine or activated charcoal washout procedure).
* Participant has received epidural, intra-articular, intramuscular, or intravenous (IV) corticosteroids during the 4 weeks prior to first administration of study drug.
* Participant has been treated with cytotoxic agents, (including but not limited to azathioprine, cyclosporine, cyclophosphamide), nitrogen mustard, chlorambucil, or other alkylating agents within 6 months prior to the first administration of the study drug.
* Participant has received or is expected to receive any live vaccinations from 3 months before first study drug administration and up to 3 months after the last study drug administration.
* Participant has received other therapeutic infectious agents within 8 weeks prior to first dose or expected to receive other therapeutic infectious agents during the study until SFU.
* Participant has received IV immunoglobulins or plasmapheresis within 6 months prior to the first administration of the study drug.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 704 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
ACR20 | Week 8 for EMA or Week 14 for FDA and NMPA
  To demonstrate the equivalence of BAT2506 and Simponi® on ACR 20 response in participants with active PsA

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital Sichuan University, Chengdu, China